CLINICAL TRIAL: NCT05353660
Title: Risk Factors of Chronic Kidney Disease-related Sarcopenia and Its Relationship With Poor Prognosis
Brief Title: Chronic Kidney Disease-related Sarcopenia With Poor Prognosis
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-122
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases; Sarcopenia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic kidney disease
  Interventions: Other: No intervention
- maintenance hemodialysis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Chronic kidney disease (CKD) has become a global public health priority over the past few decades, affecting 10-12% of the adult population and has received increasing attention. Sarcopenia describes a generalizes degenerative skeletal muscle disorder involving the loss of muscle mass, muscle function and/or physical performance. Indeed, Sarcopenia is a condition with many causes and it can be considered "primary sarcopenia" when no other cause is evident but ageing. While in the clinical practice, it also occurs in patients with chronic diseases, such as chronic kidney disease, which can be considered "secondary sarcopenia". Notably, the occurrence of sarcopenia in CKD patients is not only related with ageing, the accumulation of uremic toxins, inflammation, insulin resistance, malnutrition and oxidative stress also contribute to the muscle depletion. Moreover, sarcopenia increased risk of falls and fractures, impaired ability to perform activities of daily living, disabilities, loss of independence and increased risk of death. Hence, it is of great significance to prevent the occurrence and development of sarcopenia in patients with CKD. The purposes of this project were to investigate the prevalence of sarcopenia, further explore the risk factors for sarcopenia and detect the relationship between sarcopenia and outcomes in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.aged ≥18 years and <80 years 2.eGFR<60ml/min/1.73m2 or had received maintenance dialysis for at least 3 months.

Exclusion Criteria:

* 1.Patients with neuromuscular diseases: such as muscular dystrophy, amyotrophic lateral sclerosis, spinal cord injury, stroke, and myasthenia gravis; 2.Patients with neurodegenerative diseases: such as Alzheimer's disease, Parkinson's disease and Huntington's disease; 3.patients with advanced malignant tumors; 4.Patients with acute infectious diseases in the past 3 months; 5. Patients with serious cardiovascular or cerebrovascular disease; 6.Moderate to severe edema; 7.Patients with rheumatoid arthritis, multiple sclerosis, or acute gout that limit joint mobility; 8.Pregnant ; 9.Patients identified to be unsuitable for enrollment by the study physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from department of Nephrology, Nanfang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
sarcopenia | 1 year
  The sarcopenia is defined as: Patients with low strength: handgrip <28kg for male or <18kg for female; Or low muscle mass: appendicular skeletal muscle mass/height2 <7kg/m2 for male or <5.7kg/m2 for female; Or low performance: 6-metre walk: <1.0 m/s or 5-time chair stand test: ≥12 s
The progression of chronic kidney diseases in CKD patients | 1 year
  The progression of chronic kidney disease is defined as: Patients had a 50% or greater decrease in baseline eGFR <60 ml /min/1.73m2; Or end-stage renal disease (eGFR <15 ml /min/1.73m2, or initiation of renal replacement therapy)
All-cause mortality in maintenance hemodialysis patients | 1 year
  All-cause mortality is defined as the death due to any reasons.

SECONDARY OUTCOMES:
CVD mortality | 1 year
  CVD mortality included cerebrovascular accidents, heart failure, myocardial infarction, cardiac arrest, death caused by malignant arrhythmias, and sudden death.
cardiovascular events | 1 year
  Cardiovascular events included stroke, myocardial infarction, angina, congestive heart failure and other cardiovascular events.
Rate of participants with hospitalization. | 1 year
  Hospitalization for any reason
Rate of participants with fall. | 1 year
  Rate of participants with fall.
Rate of participants with bone fracture. | 1 year
  Rate of participants with bone fracture.
Change of quality of life | 1 year
  The quality of life is assessd by 12-item Short-Form Health Survey Questionnaire (SF-12) Survey Questionnaire (SF-12)
Frailty | 1 year
  Frailty is assessed by The FRAIL Scale. The FRAIL Scale consists of five items: fatigue, resistance, ambulation, illness, and loss of weight. The scores range from 0 to 5,with 3 to 5 as frail, 1 to 2 as pre-frail, and 0 as normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The data will be available from the corresponding author upon request, after the request is submitted and formally reviewed and approved by the Ethics Committee of Nanfang Hospital.